CLINICAL TRIAL: NCT04424589
Title: Efficacy of Myofascial Release Compared With Sham Therapy on Joint Range of Motion in Patients With Axial Spondyloarthritis.
Brief Title: Efficacy of Myofascial Release in Patients With Axial Spondyloarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPI-01-2020
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release (Experimental): Myofascial release or induction (MFR) is a widely used manual therapy treatment involving specifically guided, low-load, long-lasting mechanical forces to manipulate the myofascial complex, aimed at restoring optimal length, decreasing pain, and improving function. Manual therapists often use their hands using their knuckles, elbows, or other instrumental tools to slowly penetrate the layers of the fascia, using applied pressure with a few kilograms of force that can strain the restricted fascia, this implies a guided gentle stretch.
  The experimental group will receive 1 examination session and 6 myofascial release sessions carried out by a physiotherapist specialized in orthopedic manual therapy, superficial and deep techniques will be applied in the cervical region, for the spinal at the level of the quadratus lumborum, sacroiliac region and upper trapezius. 2 sessions per week over the course of 3 weeks.
  Interventions: Other: Myofascial release
- Sham Therapy (Sham Comparator): The control group will receive 1 examination session and 6 simulated myofascial releasesessions, where a physiotherapist will apparently apply the same techniques and maneuvers of myofascial release, however, they will not follow the basic principles of technique execution, which does a procedure with a placebo effect.
  Interventions: Other: Sham therapy

INTERVENTIONS:
Other: Myofascial release — Myofascial release or induction (IMF) is a widely used manual therapy treatment involving specifically guided, low-load, long-lasting mechanical forces to manipulate the myofascial complex, aimed at restoring optimal length, decreasing pain, and improving function. The experimental group will receive 1 examination session and 6 myofascial induction sessions carried out by a physiotherapist specialized in orthopedic manual therapy, superficial and deep techniques will be applied in the cervical region, for spinal at the level of the lumbar square, sacroiliac region and upper trapezius. 2 sessions per week over the course of 3 weeks.
  Arms: Myofascial release
Other: Sham therapy — The control group will receive 1 examination session and 6 simulated myofascial induction sessions, where a physiotherapist will apparently apply the same techniques and maneuvers of myofascial induction, however, they will not follow the basic principles of technique execution, which does a procedure with a placebo effect.
  Arms: Sham Therapy

SUMMARY:
Axial spondyloarthritis (AS), is a chronic and disabling disease that mainly affects young people, generating clear limitations in mobility and functional capacity in patients who develop this disease. Although pharmacological treatment is the basis of the therapeutic treatment of (AS), non-pharmacological treatment is a fundamental complement that guarantees the optimization of movement patterns, in turn favoring independence in the basic activities of life daily through the management and control of the derived signs and symptoms. Several studies have demonstrated the effectiveness of physiotherapy in treating symptoms in patients with AS, one of these studies is the Cochrane review developed by Dagfinrud et al. One of the techniques described by the Cochrane Review in the management of symptoms is orthopedic manual therapy (OMT), defined as a specialized area of physical therapy used for the treatment of neuro-musculoskeletal conditions, based on clinical reasoning, using approaches highly specific treatment plans that include manual techniques and therapeutic exercises.

Among these manual techniques, it includes myofascial induction as the primary technique of choice for the management of soft tissue and fascial system restrictions, it has been shown to be in rheumatic diseases such as fibromyalgia and osteoarthritis, as well as in non-inflammatory mechanical diseases such as non-specific low back pain, a low-cost, rapid therapeutic action strategy with sustained gains over time in managing global symptoms. Currently, the effects of myofascial induction on the mobility and function of patients with AS are unknown, despite the excellent results that these techniques have shown in dysfunctions of non-autoimmune musculoskeletal origin. For this reason, this study will seek to evaluate the efficacy of myofascial release compared to sham therapy in joint range of motion in patients diagnosed with axial spondyloarthritis.

DETAILED DESCRIPTION:
Trial design: Controlled parallel double blind superiority clinical trial. Participants of the trial: Patients with a diagnosis of axial spondyloarthritis, of legal age, attending the rheumatology service of an outpatient clinic in the city of Bogotá. Planned trial period: The intervention per participant is designed to develop 6 therapy sessions 2 times per week over the course of 3 weeks. It is not planned to follow up the participants in time after the end of the study and treatment time. The total duration of the project will be 4 months while the necessary population is recruited to complete the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ankylosing spondyloarthritis confirmed by rheumatologist regardless of the level of disease activity.
* Patients with cognitive ability to follow orders.
* Patients who agree to participate in the study and firm informed consent.

Exclusion Criteria:

* Patients receiving oral or parenteral coagulation therapy.
* Pregnant women
* Patients with Kinesiophobia.
* Patients with previous physical therapy in the last 15 days.
* Presence of active cancer, current treatment in chemo or radiotherapy.
* Patients who do not wish to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 3 weeks
  Index that examines 4 axial measurements (cervical rotation, Schober test, lateral trunk flexion, tragus wall distance), also includes a measurement of peripheral mobility (intermaleolar distance), The measurement of these variables is carried out comparatively, in at least two attempts, obtaining the averages of the measurements to calculate the final score based on the 11-point table.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Functional Index (BASFI) | 3 Weeks
  BASFI is a set of 10 questions designed to determine the degree of functional limitation in people with AS. The score is generated by giving a value of 1 to 10 to each of the questions, once this process has been carried out, this value is divided by 10 and the higher the score given by the scale, the greater the estimates functional limitation.
El Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 3 weeks
  This index is developed to measure disease activity in patients with ankylosing spondylitis. It consists of 6 questions that include the components of fatigue, spinal pain, joint pain / inflammation, pain in the entheses and morning stiffness. The score is generated by giving a value from 1 to 10 to each of the questions.
ASQoL (Ankylosing Spondylitis Quality of Life) | 3 Weeks
  It consists of 18 questions, with the possibility of a dichotomous answer (Yes-No) The global score ranges from 0 to 18

CONTACTS AND LOCATIONS:
Overall Officials: María Alejandra Sánchez Vera, PT, Principal Investigator — Universidad de la Sabana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perrotta FM, Musto A, Lubrano E. New Insights in Physical Therapy and Rehabilitation in Axial Spondyloarthritis: A Review. Rheumatol Ther. 2019 Dec;6(4):479-486. doi: 10.1007/s40744-019-00170-x. Epub 2019 Aug 13. PMID 31410786
- [Background] Dagfinrud H, Kvien TK, Hagen KB. The Cochrane review of physiotherapy interventions for ankylosing spondylitis. J Rheumatol. 2005 Oct;32(10):1899-906. PMID 16206344
- [Background] Cathcart E, McSweeney T, Johnston R, Young H, Edwards DJ. Immediate biomechanical, systemic, and interoceptive effects of myofascial release on the thoracic spine: A randomised controlled trial. J Bodyw Mov Ther. 2019 Jan;23(1):74-81. doi: 10.1016/j.jbmt.2018.10.006. Epub 2018 Oct 24. PMID 30691766
- [Background] Arguisuelas MD, Lison JF, Domenech-Fernandez J, Martinez-Hurtado I, Salvador Coloma P, Sanchez-Zuriaga D. Effects of myofascial release in erector spinae myoelectric activity and lumbar spine kinematics in non-specific chronic low back pain: Randomized controlled trial. Clin Biomech (Bristol). 2019 Mar;63:27-33. doi: 10.1016/j.clinbiomech.2019.02.009. Epub 2019 Feb 14. PMID 30784788
- [Result] Florez Garcia MT, Carmona L, Almodovar R, Fernandez de Las Penas C, Garcia Perez F, Perez Manzanero MA, Garcia Garcia JM, Soriano Segarra L, Jimenez Diaz JF, Mendoza Laiz N, de Miguel Mendieta E, Torre Alonso JC, Linares Ferrando LF, Collantes Estevez E, Sanz Sanz J, Zarco Montejo P. Recommendations for the prescription of physical exercise for patients with spondyloarthritis. Reumatol Clin (Engl Ed). 2019 Mar-Apr;15(2):77-83. doi: 10.1016/j.reuma.2017.06.014. Epub 2017 Aug 12. English, Spanish. PMID 28807651
- [Derived] Sanchez Vera MA, Jaimes Fernandez DA, Schleip R. Efficacy of myofascial induction compared with its simulation on joint amplitude in people with axial spondylarthritis: Protocol of a randomized controlled clinical trial. PLoS One. 2023 Oct 5;18(10):e0286885. doi: 10.1371/journal.pone.0286885. eCollection 2023. PMID 37796870